CLINICAL TRIAL: NCT00107809
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy and Safety of PROVIGIL ® (Modafinil) Treatment (100, 200, and 400 mg/Day) in Children and Adolescents With Excessive Sleepiness Associated With Obstructive Sleep Apnea/Hypopnea Syndrome
Brief Title: Study of PROVIGIL ® (Modafinil) Treatment in Children and Adolescents With Excessive Sleepiness Associated With Obstructive Sleep Apnea/Hypopnea Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1538/3028/AP/MN-OSAHS
Record Dates: First submitted 2005-04-08; First posted 2005-04-11 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Pediatric Obstructive sleep Apnea; Excessive sleepiness; CPAP; Pediatric OSAHS
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The primary objectives of the study are to determine the effectiveness of PROVIGIL treatment, compared to placebo treatment, in children and adolescents with excessive sleepiness (ES) associated with obstructive sleep apnea/hypopnea syndrome (OSAHS), as assessed by:

* mean sleep latency from the Multiple Sleep Latency Test (MSLT) (average of 4 naps performed at 0900, 1100, 1300, and 1500) at the last post baseline observation (week 6 or early termination)
* the Clinical Global Impression of Change (CGI-C) ratings for ES, at the last post baseline observation (week 6 or early termination).

DETAILED DESCRIPTION:
PROVIGIL is a trademark of Genelco, SA, licensed to Cephalon, Inc.

ELIGIBILITY:
Inclusion Criteria:

* A boy or girl aged 6 through 16 years, inclusive
* Meet the minimal criteria established by the International Classification of Sleep Disorders (ICSD) manual of the American Academy of Sleep Medicine (AASM) for OSAHS as assessed by all of the following: *clinical history;

  *have a previous diagnosis of OSAHS on the basis of NPSG (nocturnal polysomnogram) and/or MSLT at any time before the screening visit. If the patient is a current user of CPAP (continuous positive airway pressure) therapy and is appropriately titrated on CPAP, the AHI ≥5 inclusion criterion is not applicable; *NPSG (nocturnal polysomnogram) (as evaluated by the investigator) to rule out other sleep disorders (ie, narcolepsy and periodic limb movement with sleep [PLMs]).
* Have ES (CGI-S [Clinical Global Impression of Severity] ≥4) that is not a direct result of inadequate sleep hygiene or other medical disorder
* Are in good health as determined by a medical and psychiatric history, physical examination, ECG, and clinical laboratory tests
* For patients who are not current users of CPAP therapy or who are not appropriately titrated on CPAP: have an average of 5 or more apneic/hypopneic episodes per hour of nocturnal sleep, as assessed by the NPSG at the baseline visit (AHI [apnea/hypopnea index] ≥5)
* Are currently users of CPAP therapy or have tried and not tolerated the current standards of care for OSAHS and continue to have residual sleepiness (ie, patients who comply with CPAP use, patients who are unable to tolerate or comply with CPAP therapy, patients who have had surgical removal of tonsils and adenoids or for whom this surgery is not warranted, and patients who have attempted or are on an ongoing weight loss program)
* Have an O2 saturation of at least 85%, based on the investigator's assessment of the patient's health
* Have blood pressure values greater than those for the 5th percentile and less than the 95th percentile for age on the National High Blood Pressure Education Program guidelines for blood pressure levels for boys and girls ages 6 through 16 years
* Girls who are post menarche or sexually active must have a negative urine pregnancy test prior to the baseline visit, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implanted, or injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence.
* Be able to swallow a placebo tablet the same size and shape as the study drug tablet
* Negative UDS (urine drug screen) for any illicit drug, alcohol (ethanol), stimulants, or modafinil at screening; if positive for stimulants or modafinil (prescribed for ES) at the screening visit, UDS to be repeated after washout period and before the baseline visit
* Have a parent or legal guardian who is willing to participate in the study

Exclusion Criteria:

* Have any other disorder(s) that could be considered the primary cause of ES (eg, self induced sleep deprivation)
* Have a past or present seizure disorder (except history of a single febrile seizure), a history of psychosis, or of clinically significant head trauma (eg, brain damage) or past neurosurgery
* Have periodic limb movement (PLM) arousal index greater than 5 (ie, >5 PLMs with arousals per hour of sleep)
* Have a history of suicide attempt, or are at suicidal risk
* A clinically significant drug sensitivity to stimulants such as amphetamine, dextroamphetamine, methylphenidate, or pemoline; and/or modafinil or any of its components
* Use of any prescription (eg, clonidine, guanfacine) or nonprescription (over the counter [OTC]) medications, including dietary supplements with psychoactive properties (eg, any OTC medications or supplements containing ephedrine [ie, ma huang or ephedra], pseudoephedrine, caffeine, or phenylpropanolamine) or sedating properties (ie, antihistamines or sedative hypnotics) within 1 week of the baseline visit
* Use of any MAO (monoamine oxidase) inhibitors or SSRIs (selective serotonin reuptake inhibitors) within 2 weeks of the baseline visit
* Received any investigational drug (except modafinil) within 4 weeks of the baseline visit
* Any disorder that could interfere with drug absorption, distribution, metabolism, or excretion (including previous gastrointestinal surgery)
* Active, clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other major clinically significant disorder/disease
* Any clinically significant deviation from the normal range(s) in the physical examination or ECG findings, or clinical laboratory test results (ie, serum chemistry, hematology, and urinalysis) at the screening or baseline visit
* ANC (absolute neutrophil count) below the lower limit of normal at the screening visit (NOTE: If the ANC is below the lower limit of normal at the baseline visit, the medical monitor will be consulted for continued eligibility in the study.)
* Seated pulse outside the range of 60 through 115 bpm after resting for 5 minutes
* A history of alcohol, narcotic, or any other substance abuse or dependence as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM IV) criteria
* A total daily intake of more than 250 mg of caffeine per day (eg, approximately five 12 ounce caffeinated sodas, 2.5 cups of coffee or tea, or about 12.5 ounces of chocolate per day) within 1 week of the baseline visit
* Pregnant or lactating/nursing girl; any girl who becomes pregnant during the study will be withdrawn
* A clinically significant illness within 4 weeks of the baseline visit; or is symptomatic for any clinically significant illness at the screening or baseline visit.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140
Dates: Start 2004-10; Study Completion 2005-09

PRIMARY OUTCOMES:
Mean sleep latency from the Multiple Sleep Latency Test (MSLT) (average of 4 naps performed at 0900, 1100, 1300, and 1500) at the last post baseline observation (week 6 or early termination)
The Clinical Global Impression of Change (CGI-C) ratings for ES, at the last post baseline observation (week 6 or early termination)

SECONDARY OUTCOMES:
The Clinical Global Impression of Change (CGI-C) ratings for severity of ES
The total score from the Pediatric Daytime Sleepiness Scale (PDSS)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (60):
  - Robert Doekel, Jr., M.D., Birmingham, Alabama
  - Derek Loewy, Ph.D., Tucson, Arizona
  - Stuart Quan, M.D., Tucson, Arizona
  - Joseph McCarty, M.D., Fort Smith, Arkansas
  - John L. Carroll, M.D., Little Rock, Arkansas
  - Julie Thompson-Dobkin, D.O., Huntington Beach, California
  - Mark Buchfuhrer, M.D., Long Beach, California
  - Yury Furman, M.D., Los Angeles, California
  - Stuart Menn, M.D., Palm Springs, California
  - Richard Shubin, M.D., Pasadena, California
  - Lawrence Sher, M.D., Rolling Hills Estates, California
  - Milton K. Erman, M.D., San Diego, California
  - Stephen Brooks, M.D., San Francisco, California
  - Paul Haberman, M.D., Santa Monica, California
  - Jed Black, M.D., Stanford, California
  - Amerigo Padilla, M.D., Miami, Florida
  - Martin A. Cohn, M.D., Naples, Florida
  - D. Alan Lankford, Ph.D., Atlanta, Georgia
  - Gary Montgomery, M.D., Atlanta, Georgia
  - Jerry Silverboard, M.D., Atlanta, Georgia
  - Stephen H. Sheldon, D.O., FAAP, Chicago, Illinois
  - Michael Kohrman, M.D., Chicago, Illinois
  - Anna Ivanenko, M.D., Ph.D., Maywood, Illinois
  - Henry Lahmeyer, M.D., Northfield, Illinois
  - James Cook, M.D., Danville, Indiana
  - William Leeds, D.O., Topeka, Kansas
  - Karen Waters, M.D., Louisville, Kentucky
  - Margaret Ann Springer, M.D., Shreveport, Louisiana
  - Helene A. Emsellem, M.D., Chevy Chase, Maryland
  - Marc Raphaelson, M.D., Frederick, Maryland
  - Daniela Minecan, M.D., Ann Arbor, Michigan
  - George Zureikat, M.D., Flint, Michigan
  - Pradeep Sahota, M.D., Columbia, Missouri
  - William Torch, M.D., MS, Reno, Nevada
  - Kathleen Ryan, M.D., Mount Laurel, New Jersey
  - Sushmita Mikkilineni, M.D., New Brunswick, New Jersey
  - Monroe Karetzky, M.D., Newark, New Jersey
  - Lee Brooks, M.D., Princeton, New Jersey
  - Marc Seelagy, M.D., Trenton, New Jersey
  - Gary Zammit, M.D., New York, New York
  - James Lee, M.D., Charlotte, North Carolina
  - Raouf Amin, MD, Cincinnati, Ohio
  - Martin Scharf, Ph.D., Cincinnati, Ohio
  - Markus H. Schmidt, M.D., Ph.D., Dublin, Ohio
  - Michael Neeb, Ph.D., Toledo, Ohio
  - William C. Orr, Ph.D., Oklahoma City, Oklahoma
  - Jorg Pahl, M.D., Oklahoma City, Oklahoma
  - Dainis Irbe, M.D., Eugene, Oregon
  - William Pistone, M.D., Allentown, Pennsylvania
  - Jeffery Gould, M.D., Bethlehem, Pennsylvania
  - Guillermo Borrero, M.D., Clairton, Pennsylvania
  - Judith Owens, M.D., MPH, Providence, Rhode Island
  - Richard Bogan, M.D., FCCP, Columbia, South Carolina
  - Julie Jacques, D.O., Morristown, Tennessee
  - John Hudson, M.D., Austin, Texas
  - David Sperry, M.D., Dallas, Texas
  - Todd J. Swick, M.D., Houston, Texas
  - Jerry J. Tomasovic, M.D., San Antonio, Texas
  - James M. Ferguson, M.D., Salt Lake City, Utah
  - Ralph A. Pascualy, M.D., Seattle, Washington
- Canada (4):
  - Adam Moscovitch, M.D., Calgary, Alberta
  - Leonid Kayumov, M.D., Scarborough Village, Ontario
  - Mortimer Mamelak, M.D., Toronto, Ontario
  - Allen Denys, M.D., Windsor, Ontario